CLINICAL TRIAL: NCT04706689
Title: The Development and Validation of the SWADOC Tool: A Study Protocol for a Multicentric Prospective Cohort Study
Brief Title: Development and Validation of the SWADOC Tool
Status: Recruiting | Type: Observational
Sponsor: University of Liege (Other)
Collaborators: Centre du Cerveau², Centre hospitalier universitaire de Liège (Unknown); Centre de Traumatologie et de Réadaptation de Jette (Erasme, ULB) (Unknown); Cliniques de Soins Spécialisés Valdor-Pèrî (Unknown); Centre Hospitalier Neurologique William Lennox (UCL) (Unknown); Centre Hospitalier Universitaire de Liege (Other); Centre Hospitalier Universitaire de Nīmes (Other); Uzès hospital (Unknown); Fontfroide functional re-education centre, Montpellier, France (Unknown)
Responsible Party: Principal Investigator, Olivia Gosseries, Neuropsychologist, PhD, Co-director of the Coma Science Group, Research Associate at FRS-FNRS, University of Liege
Other Study IDs: 2020_79
Record Dates: First submitted 2021-01-07; First posted 2021-01-13 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Swallowing Disorders; Dysphagia; Disorders of Consciousness; Assessment Tool; Speech Therapy
Keywords: swallowing; dysphagia; disorders of consciousness; severe brain injury
MeSH Terms: conditions — Deglutition Disorders; Consciousness Disorders; Communication Disorders; Brain Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Unresponsive wakefulness syndrome patients (UWS): The level of consciousness will be assessed with the Simplified Evaluation of CONsciousness Disorder (SECONDs) and the Coma Recovery Scale-Revised (CRS-R).
  Interventions: Behavioral: SWADOC tool; Behavioral: FOTT-SAS
- Minimally conscious patients MINUS (MCS-): The level of consciousness will be assessed with the Simplified Evaluation of CONsciousness Disorder (SECONDs) and the Coma Recovery Scale-Revised (CRS-R).
  Interventions: Behavioral: SWADOC tool; Behavioral: FOTT-SAS
- Minimally conscious patients PLUS: The level of consciousness will be assessed with the Simplified Evaluation of CONsciousness Disorder (SECONDs) and the Coma Recovery Scale-Revised (CRS-R).
  Interventions: Behavioral: SWADOC tool; Behavioral: FOTT-SAS
- Patients emerging from the minimally conscious state (EMCS): The level of consciousness will be assessed with the Simplified Evaluation of CONsciousness Disorder (SECONDs) and the Coma Recovery Scale-Revised (CRS-R).
  Interventions: Behavioral: SWADOC tool; Behavioral: FOTT-SAS

INTERVENTIONS:
Behavioral: SWADOC tool — The tool explores some oral and pharyngeal components of swallowing as well as a range of prerequisite and related components of swallowing in DOC patients.
  It is composed of an average of 50 qualitative items and a subsection named "SWADOC-scored" comprising 8 quantitative items.
Behavioral: FOTT-SAS — Facial Oral Tract Therapy Swallowing Assessment of Saliva : the results of the SWADOC-scored in one of the sessions will be compared to the FOTT Swallowing Assessment of Saliva (FOTT-SAS) (27). The test is based on 7 questions under which if items 1-4 are answered "Yes" and items 5-7 are answered "No", oral intake should be initiated. The FOTT-SAS includes items that can be scored based on the administration of the SWADOC tool. In that respect, no additional administration will be required

SUMMARY:
Background: After a period of coma, patients with severe brain injury may present disorders of consciousness (DOC). A wide proportion of these patients also suffer from severe dysphagia. Assessment and therapy of swallowing disabilities of DOC patients are essential because dysphagia has major functional consequences and comorbidities. Dysphagia evaluation in patients with DOC is hampered by the lack of adapted tools. The first aim of the study was to develop a new tool, the SWallowing Assessment in Disorders Of Consciousness (SWADOC), and propose a validation protocol. The SWADOC tool has been developed to help therapists to apprehend components related to swallowing in patients with DOC. The second aim is to appreciate the relationship between patients' level of consciousness and SWADOC items and scores.

Method/design: In this multicentric prospective cohort, 104 patients with DOC will be tested three times during two consecutive days with the SWADOC tool. Statistical analyses will focus on the reliability and validity of the SWADOC tool, especially the intra and inter-rater reliability, internal consistency, measures of dispersion and concurrent validity with the FOTT Swallowing Assessment of Saliva (FOTT-SAS). The level of consciousness will be assessed with the Simplified Evaluation of CONsciousness Disorders (SECONDs) and the Coma Recovery Scale-Revised (CRS-R)

Discussion: The assessment of swallowing abilities among patients with DOC is the first necessary step towards the development of an individualized dysphagia care plan. A validated scoring tool will be essential for clinicians to better apprehend dysphagia in DOC patients and to document the evolution of their disorders.

ELIGIBILITY:
Inclusion Criteria :

* Age above 18-year-old
* Perfect knowledge of French language before the injury
* Previous event of coma phase caused by a severe acquired brain injury
* Medical stability (absence of mechanical ventilation and sedation, no acute medical pathology such as infection or respiratory distress)
* No neurological or otorhinolaryngological disease which can impact swallowing prior to the brain injury
* Minimum of 28 days since the acquired brain injury at inclusion
* Diagnosis of UWS, MCS-, MCS+ or EMCS based on the CRS-R or SECONDs
* Informed consent from legal representative of the patient
* Affiliated patient or beneficiary of a health insurance plan (for French participants only).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will be carried out in patients with DOC or emerging from DOC following severe acquired brain injury. Patients will be divided into four groups according to their clinical diagnosis assessed with the Simplified Evaluation of CONsciousness Disorders (SECONDs): UWS, MCS-, MCS+ and EMCS. Participants will be recruited from inpatient neurological rehabilitation programs in post-coma units and rehabilitation services, or hospitalized for an evaluation of multimodal assessment of consciousness for diagnostic and prognostic purposes.
  We will include 26 patients in each group, which will result in a total of 104 patients.
Sampling Method: Non-Probability Sample
Enrollment: 104 (Estimated)
Dates: Start 2020-07-24 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in the SWADOC-scored during three sessions (Examiner 1) - Intra-reliability | 15-25 minutes (3 times in 5 business days)
  The SWallowing Assessment in Disorders Of Consciousness (SWADOC) tool is composed of an average of 50 qualitative and quantitative items. The subsection "SWADOC-scored" includes the 8 quantitative items. Four items are linked to the oral phase and four to the pharyngeal phase. For each quantitative item, patient's abilities are rated on a four-level severity scale ranging from 0 to 3. These levels correspond to item scores that can be added together to calculate 3 performance scores: the oral phase sub-score (sum of the 4 oral item scores - minimum of 0, maximum of 12), the pharyngeal phase sub-score (sum of the 4 pharyngeal item scores - minimum of 0, maximum of 12) and the total swallowing score (sum of the 8 item scores - minimum of 0, maximum of 24).
  The better the score is, the better the swallowing is.
SECONDs | 7 minutes (immediately before or after the SWADOC tool in each of the three sessions)
  The Simplified Evaluation of CONsciousness Disorders (SECONDs): it features a shorter administration time (median of 7 minutes) and required only a mirror as material. It consists of 8 items: observation and reporting spontaneous behaviors, response to command, communication, visual pursuit and fixation, pain localization, oriented behaviors and arousal. The SECONDs provides a total score directly reflecting one diagnosis (0 = coma, 1 = UWS, 2-5 = MCS-, 6-7 = MCS+, 8 = EMCS). The better the score is, the better the consciousness level is.

SECONDARY OUTCOMES:
SWADOC-scored by Examiner 2 (inter-reliability) | 15-25 minutes - immediately before or after one of the three sessions
  The SWallowing Assessment in Disorders Of Consciousness (SWADOC) tool is composed of an average of 50 qualitative and quantitative items. The subsection "SWADOC-scored" includes the 8 quantitative items. Four items are linked to the oral phase and four to the pharyngeal phase. For each quantitative item, patient's abilities are rated on a four-level severity scale ranging from 0 to 3. These levels correspond to item scores that can be added together to calculate 3 performance scores: the oral phase sub-score (sum of the 4 oral item scores - minimum of 0, maximum of 12), the pharyngeal phase sub-score (sum of the 4 pharyngeal item scores - minimum of 0, maximum of 12) and the total swallowing score (sum of the 8 item scores - minimum of 0, maximum of 24). The better the score is, the better the swallowing is.
FOTT-SAS (Examiner 1) | Immediately after one of the three sessions
  FOTT-SAS (Facial Oral Tract Therapy Swallowing Assessment of Saliva) The FOTT-SAS is a reliable assessment for detecting aspiration risk in patients with acquired brain injury.
  The test is based on 7 questions under which if items 1-4 are answered "Yes" and items 5-7 are answered "No", oral intake should be initiated (the better the score is, the better the swallowing is, minimum of 0, maximum of 7).
  The observations made during the assessment will permit to score the FOTT-SAS and verify the concurrent validity of the SWADOC tool.

CONTACTS AND LOCATIONS:
Overall Officials: Olivia Gosseries, PhD, Study Director — University of Liege, Giga Consciousness
Locations (8):
- Belgium (5):
  - Centre Hospitalier Neurologique William Lennox (UCL), Ottignies-Louvain-la-Neuve, Brabant Wallon
  - Centre neurologique et de réadaptation fonctionnelle de Fraiture-en-Condroz, Fraiture
  - Centre de Traumatologie et de Réadaptation de Jette (Erasme, ULB), Jette
  - Centre du Cerveau², University Hospital of Liège, Liège
  - Cliniques de Soins Spécialisés Valdor-Pèrî, Liège
- France (3):
  - Fontfroide functional re-education centre, Montpellier
  - CHU Nîmes, Nîmes
  - Uzès hospital, Uzès

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Melotte E, Maudoux A, Delhalle S, Lagier A, Thibaut A, Aubinet C, Kaux JF, Vanhaudenhuyse A, Ledoux D, Laureys S, Gosseries O. Swallowing in individuals with disorders of consciousness: A cohort study. Ann Phys Rehabil Med. 2021 Jul;64(4):101403. doi: 10.1016/j.rehab.2020.04.008. Epub 2020 Jul 18. PMID 32535170
- [Background] Sanz LRD, Aubinet C, Cassol H, Bodart O, Wannez S, Bonin EAC, Barra A, Lejeune N, Martial C, Chatelle C, Ledoux D, Laureys S, Thibaut A, Gosseries O. SECONDs Administration Guidelines: A Fast Tool to Assess Consciousness in Brain-injured Patients. J Vis Exp. 2021 Feb 6;(168). doi: 10.3791/61968. PMID 33616111
- [Background] Mortensen J, Jensen D, Kjaersgaard A. A validation study of the Facial-Oral Tract Therapy Swallowing Assessment of Saliva. Clin Rehabil. 2016 Apr;30(4):410-5. doi: 10.1177/0269215515584381. Epub 2015 Apr 28. PMID 25920675
- [Background] Bicego A, Lejoly K, Maudoux A, Lefebvre P, Laureys S, Schweizer V, Diserens K, Faymonville ME, Vanhaudenhuyse A. [Swallowing in disorders of consciousness]. Rev Neurol (Paris). 2014 Oct;170(10):630-41. doi: 10.1016/j.neurol.2014.04.004. Epub 2014 Jun 18. French. PMID 24952924
- [Background] Wannez S, Gosseries O, Azzolini D, Martial C, Cassol H, Aubinet C, Annen J, Martens G, Bodart O, Heine L, Charland-Verville V, Thibaut A, Chatelle C, Vanhaudenhuyse A, Demertzi A, Schnakers C, Donneau AF, Laureys S. Prevalence of coma-recovery scale-revised signs of consciousness in patients in minimally conscious state. Neuropsychol Rehabil. 2018 Dec;28(8):1350-1359. doi: 10.1080/09602011.2017.1310656. Epub 2017 Apr 11. PMID 28399715
- [Derived] Melotte E, Belorgeot M, Herr R, Simon J, Kaux JF, Laureys S, Sanz LRD, Lagier A, Morsomme D, Pellas F, Gosseries O. The Development and Validation of the SWADOC: A Study Protocol for a Multicenter Prospective Cohort Study. Front Neurol. 2021 Apr 29;12:662634. doi: 10.3389/fneur.2021.662634. eCollection 2021. PMID 33995257